CLINICAL TRIAL: NCT06111586
Title: A 52-week Randomized, Double-blind, Placebo-controlled, Multi-center Phase 2b Study With a 52-week Blinded Extension and an Optional Open-label Extension - Assessing Safety and Efficacy of Frexalimab, a CD40L-antagonist Monoclonal Antibody, for Preservation of Pancreatic β-cell Function in Adults and Adolescents With Newly Diagnosed Type 1 Diabetes on Insulin Therapy
Brief Title: FrexalimAB in Preservation of Endogenous insULIN Secretion Compared to Placebo in adUlts and Adolescents on Top of inSulin Therapy (FABULINUS)
Acronym: FABULINUS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRI17476; U1111-1275-9618 (Registry Identifier: ICTRP); 2022-500531-36 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Frexalimab Dose 1 (Experimental)
  Interventions: Drug: Frexalimab; Drug: Insulin
- Frexalimab Dose 2 (Experimental)
  Interventions: Drug: Frexalimab; Drug: Insulin
- Frexalimab Dose 3 (Experimental)
  Interventions: Drug: Frexalimab; Drug: Insulin
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo; Drug: Insulin

INTERVENTIONS:
Drug: Frexalimab — Intravenous (IV) Infusion at Day 1 and subcutaneous (SC) Injection from W2 to W102
  Arms: Frexalimab Dose 1; Frexalimab Dose 2; Frexalimab Dose 3
Drug: Placebo — IV Infusion at Day 1 and SC Injection from W2 to W102
  Arms: Placebo
Drug: Insulin — SC injection, dose and frequency will be established and/or adjusted by investigator

SUMMARY:
This is a randomized, parallel group, double-blind Phase 2 study with a 52-week blinded extension evaluating the safety and efficacy of 3 dose levels of frexalimab in comparison with placebo in participants with newly diagnosed T1D on insulin treatment.

Study details include:

Screening period: at least 3 weeks and up to 5 weeks

Double-blind treatment period (104 weeks):

* Main treatment period: 52 weeks
* Blinded extension: 52 weeks Optional Open Label Extension: 104 weeks Safety follow-up: up to 26 weeks The treatment duration will be up to 104 weeks, the total study duration will be up to 135 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet the criteria of T1D according to American Diabetes Association
* Initiated exogenous insulin replacement therapy not longer than 90 days prior to screening visit at which random C-peptide will be assessed (V1).
* Receiving at least one of the following T1D standard of care (SOC), insulin hormone replacement therapy

  * one or multiple daily injections (MDI) of basal insulin, prandial insulin and/or premixed insulin, or
  * continuous subcutaneous insulin infusion (CSII)
* Participants must be positive for at least 1 of the following T1D autoantibodies confirmed by medical history and/or obtained at study screening:

  * Glutamic acid decarboxylase (GAD-65)
  * Insulinoma Antigen-2 (IA-2)
  * Zinc-transporter 8 (ZnT8) or
  * Insulin (if obtained not later than 10 days after exogenous insulin therapy initiation)
* Have random C-peptide levels ≥ 0.2 nmol/L determined at screening visit.
* Be vaccinated according to the local vaccination schedule. Any vaccinations should take place at least 28 days prior to randomization for non-live vaccines and at least 3 months prior to randomization for live vaccines.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

Exclusion Criteria:

* Serious systemic viral, bacterial or fungal infection (eg, pneumonia, pyelonephritis), infection requiring hospitalization or IV antibiotics or significant chronic viral (including history of recurrent or active herpes zoster, acute or active cytomegalovirus (CMV), Epstein-Barr Virus (EBV) as determined at screening), bacterial, or fungal infection (eg, osteomyelitis) 30 days before and during screening.
* Participants with a history of invasive opportunistic infections, such as, but not limited to histoplasmosis, listeriosis, coccidioidomycosis, candidiasis, pneumocystis jirovecii, and aspergillosis, regardless of resolution.
* Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, chest X-rays (posterior anterior and lateral), and/or TB testing. Blood testing (eg, QuantiFERON® TB Gold test) is strongly preferred; if not available, any local approved TB test is allowed.
* Evidence of any clinically significant, severe or unstable, acute or chronically progressive, uncontrolled infection, medical or surgical condition (eg, but not limited to, cerebral, cardiac, pulmonary, renal, hepatic, gastrointestinal, neurologic, acquired or inherited bone/skeletal disorders including repeated bone fractures for unknown reason, juvenile osteoporosis, osteogenesis imperfecta, osteochondropathies, or any known immune deficiency), or any condition that may affect participant safety in the judgment of the Investigator (including vaccinations which are not updated based on local regulation).
* History or current hypogammaglobulinemia.
* History of a systemic hypersensitivity reaction or significant allergies, other than localized injection site reaction, to any humanized mAb. Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear IgA dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* Has other autoimmune diseases (eg, rheumatoid arthritis [RA], polyarticular juvenile idiopathic arthritis [pJIA], psoriatic arthritis [PsA], ankylosing spondylitis [AS], MS, SLE), that require treatment with biologic drugs (mono or polyclonal antibodies) or systemic corticosteroid therapy (at discretion of investigator).
* History, clinical evidence, suspicion or significant risk for thromboembolic events, as well as myocardial infarction, stroke, antiphospholipid syndrome, other prothrombotic disorders and/or participants requiring antithrombotic treatment.
* Diabetes of forms other than autoimmune T1D that include but is not limited to genetic forms of diabetes, maturity-onset diabetes of the young (MODY), latent autoimmune diabetes of the adult (LADA), secondary to medications or surgery, type 2 diabetes by judgement of the investigator.
* History of malignancy of any organ system, treated or untreated, within 5 years of screening, regardless of whether there is evidence of local recurrence or metastases.
* Systemic corticosteroids (duration > 7 days), adrenocorticotropic hormone 1 month prior to screening.
* Any IV, IM or SC administered biologic treatments, < 3 months or < than 5 half-lives (whichever is longer), prior to randomization.
* Any live (attenuated or viral-vector) vaccine (including but not limited to varicella zoster, oral polio, nasal influenza, rabies) within 3 months prior to randomization.
* Any non-live (inactivated, mRNA, recombinant, conjugate, toxoid) vaccine administered less than 28 days prior to randomization.
* Other medications not compatible or interfering with IMP at discretion of investigator.
* Any immunosuppressive therapy within 12 weeks prior to randomization.
* Course of Thymoglobulin®, teplizumab or other immunomodulatory treatments at any time.
* Any drugs that may be used for treatment of T1D and type 2 diabetes other than insulin including but not limited to metformin, glucagon-like peptide 1 (GLP-1) agonists and sodium-glucose co-transporter-2 and 1 (SGLT2/1) inhibitor and verapamil within 2 weeks prior to screening.
* Abnormal laboratory test(s) at screening.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2027-04-28 (Estimated); Study Completion 2030-10-29 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to W52 in mean 2h mixed meal tolerance test (MMTT) stimulated C-peptide concentration | Baseline to Week 52
  mixed meal tolerance test (MMTT) stimulated C-peptide concentration is to be calculated from AUC

SECONDARY OUTCOMES:
Time in range (70-180 mg/dL), assessed by CGM at W52 and W104 | At Week 52 and Week 104
Proportion of participants who remain C-peptide positive (mean 2h MMTT stimulated C-peptide concentration ≥0.2 nmol/L) at W52 and W104 | At Week 52 and Week 104
  mixed meal tolerance test (MMTT) stimulated C-peptide concentration is to be calculated from AUC
Proportion of participants with reduction from baseline to W52 and W104 of less than 10% in mean 2h MMTT stimulated C-peptide concentration | From baseline to Week 52 and Week 104
  mixed meal tolerance test (MMTT) stimulated C-peptide concentration is to be calculated from AUC
Proportion of participants with partial remission at W52 and W104 (defined as IDAA1c score ≤9.0, where it is calculated as HbA1c [%] + 4x insulin dose [IU/kg/day]) | At Week 52 and Week 104
Change from baseline to W52 and W104 in insulin dose [IU/kg/day] | From baseline to Week 52 and Week 104
HbA1c level and its change from baseline at W52 and W104 | From baseline to Week 52 and Week 104
Proportion of participants with HbA1c ≤6.5% and requiring no injections of exogenous insulin at W52 and W104 | At Week 52 and Week 104
Proportion of participants with HbA1c ≤6.5% and requiring ≤0.25 IU of insulin at W52 and W104 | At Week 52 and Week 104
Proportion of participants with HbA1c <7% at W52 and W104 | At Week 52 and Week 104
Incidence of treatment emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs) and TEAEs leading to treatment discontinuation | Until Week 130
Number of participants with at least one hypoglycemic event | Until Week 130
Number of participants with at least one hyperglycemic episode | Until Week 130
Number of participants with at least one diabetic ketoacidosis (DKA) event | Until Week 130
Number of participants with clinically significant changes in vital signs, electrocardiogram (ECG), and/or laboratory evaluation | Until Week 130
Height and growth rate over time (for participants <18 y.o. at screening) | Until Week 130
Frexalimab plasma concentrations over time | Until Week 104
Incidence of anti-drug antibodies (ADAs) over time | Until Week 130
Change from baseline to W52 and W104 in PedsQL Diabetes Symptoms domain score (all participants) | From baseline to Week 52 and Week 104
Change from baseline to W52 and W104 in Pediatric Quality of Life (PedsQL) Diabetes Management domain score (all participants) | From baseline to Week 52 and Week 104
Change from baseline to W52 and W104 in Problem Areas In Diabetes (PAID) total score (all participants) | From baseline to Week 52 and Week 104
Change from baseline to W52 and W104 in Diabetes Treatment Satisfaction Questionnaires (DTSQs) total and item scores (all participants) | From baseline to Week 52 and Week 104
Change from baseline to W52 and W104 in PAID immediate and theoretical domain scores (caregivers of all participants 12-17 y.o.) | From baseline to Week 52 and Week 104
Change from baseline to W52 and W104 in DTSQs Total and item scores (caregivers of all participants 12-17 y.o.) | From baseline to Week 52 and Week 104
Time in tight range (TITR, 70 - 140 mg/dL), assessed by CGM at W52 and W104 | Time in tight range (TITR, 70 - 140 mg/dL), assessed by CGM at W52 and W104
Change from baseline to W104 in mean 2h mixed meal tolerance test (MMTT) stimulated C-peptide concentration, calculated from AUC | From baseline to Week 104
Change from baseline to W52 in IDAA1c score | From baseline to Week 52

CONTACTS AND LOCATIONS:
Locations (79):
- United States (14):
  - University of California San Francisco - Mission Bay- Site Number : 8400012, San Francisco, California
  - University of Colorado - Anschutz Medical Campus- Site Number : 8400003, Aurora, Colorado
  - University of Florida College of Medicine- Site Number : 8400010, Gainesville, Florida
  - University of Miami Hospital- Site Number : 8400013, Miami, Florida
  - AdventHealth Orlando- Site Number : 8400002, Orlando, Florida
  - Rocky Mountain Diabetes and Osteoporosis Center- Site Number : 8400009, Idaho Falls, Idaho
  - NorthShore University Health System - Endeavor Health Medical Group - Skokie - Woods Drive- Site Number : 8400007, Skokie, Illinois
  - Joslin Diabetes Center - Boston- Site Number : 8400015, Boston, Massachusetts
  - University at Buffalo - Downtown Campus- Site Number : 8400004, Buffalo, New York
  - University of North Carolina at Chapel Hill- Site Number : 8400001, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center- Site Number : 8400019, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia Site Number : 8400005, Philadelphia, Pennsylvania
  - University of Texas - Southwestern Medical Center- Site Number : 8400011, Dallas, Texas
  - Benaroya Research Institute at Virginia Mason- Site Number : 8400016, Seattle, Washington
- Austria (2):
  - Investigational Site Number : 0400004, Linz
  - Investigational Site Number : 0400001, Vienna
- Belgium (2):
  - Investigational Site Number : 0560002, Brussels
  - Investigational Site Number : 0560001, Leuven
- Canada (5):
  - Investigational Site Number : 1240001, Vancouver, British Columbia
  - Investigational Site Number : 1240007, London, Ontario
  - Investigational Site Number : 1240005, Montreal, Quebec
  - Investigational Site Number : 1240004, Montreal, Quebec
  - Investigational Site Number : 1240003, Montreal, Quebec
- Czechia (3):
  - Investigational Site Number : 2030003, Ostrava
  - Investigational Site Number : 2030002, Prague
  - Investigational Site Number : 2030001, Prague
- Investigational Site Number : 2080005, Herlev, Denmark
- Finland (4):
  - Investigational Site Number : 2460001, Helsinki
  - Investigational Site Number : 2460004, Oulu
  - Investigational Site Number : 2460003, Tampere
  - Investigational Site Number : 2460002, Turku
- France (5):
  - Investigational Site Number : 2500004, Corbeil-Essonnes
  - Investigational Site Number : 2500005, Mont-de-Marsan
  - Investigational Site Number : 2500006, Paris
  - Investigational Site Number : 2500007, Pontoise
  - Investigational Site Number : 2500003, Saint-Herblain
- Germany (4):
  - Investigational Site Number : 2760003, Dresden
  - Investigational Site Number : 2760001, Hanover
  - Investigational Site Number : 2760002, Oldenburg in Holstein
  - Investigational Site Number : 2760004, Ulm
- Hungary (5):
  - Investigational Site Number : 3480001, Balatonfüred
  - Investigational Site Number : 3480004, Budapest
  - Investigational Site Number : 3480002, Nyíregyháza
  - Investigational Site Number : 3480003, Nyíregyháza
  - Investigational Site Number : 3480006, Székesfehérvár
- Italy (8):
  - AOU delle Marche - Ospedale G. Salesi-Site Number : 3800008, Torrette, Ancona
  - Azienda Ospedaliera Universitaria Meyer IRCCS-Site Number : 3800003, Florence, Firenze
  - IRCCS Ospedale San Raffaele-Site Number : 3800006, Milan, Milano
  - Azienda Ospedaliera Universitaria 'Federico II'-Site Number : 3800009, Naples, Napoli
  - Ospedale Pediatrico Bambin Gesu IRCCS-Site Number : 3800007, Rome, Roma
  - Azienda Ospedaliero-Universitaria Maggiore Della Carità-Site Number : 3800001, Novara
  - Azienda Socio Sanitaria Territoriale Dei Sette Laghi - Ospedale Filippo del Ponte-Site Number : 3800002, Varese
  - Azienda Ospedaliera Universitaria Integrata Verona - Centro regionale di Diabetologia Pediatrica-Site Number : 3800004, Verona
- Poland (8):
  - Investigational Site Number : 6160006, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160004, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160001, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160007, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160008, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6160002, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160009, Szczecin, West Pomeranian Voivodeship
  - Investigational Site Number : 6160005, Lodz
- Investigational Site Number : 7050001, Ljubljana, Slovenia
- Spain (7):
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240002, Esplugues de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240005, Oviedo, Principality of Asturias
  - Investigational Site Number : 7240003, Seville, Sevilla
  - Investigational Site Number : 7240004, Málaga
  - Investigational Site Number : 7240006, Valencia
  - Investigational Site Number : 7240007, Vitoria-Gasteiz, Álava
- Sweden (3):
  - Investigational Site Number : 7520002, Solna
  - Investigational Site Number : 7520001, Stockholm
  - Investigational Site Number : 7520003, Stockholm
- United Kingdom (7):
  - Investigational Site Number : 8260001, Cambridge, Cambridgeshire
  - Investigational Site Number : 8260009, Dundee, Dundee City
  - Investigational Site Number : 8260003, Birmingham, England
  - Investigational Site Number : 8260007, Birmingham, England
  - Investigational Site Number : 8260010, Glasgow, Glasgow City
  - Investigational Site Number : 8260004, Leicester, Leicestershire
  - Investigational Site Number : 8260006, Harrow, London, City of

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DRI17476 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25574&tenant=MT_SNY_9011